CLINICAL TRIAL: NCT04773483
Title: Quorn in Community Health Experiment
Acronym: QUICHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Marlow Foods Ltd (Unknown); NIHR Exeter Clinical Research Facility (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201021-B-02 Wall
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quorn Food products (Active Comparator)
  Interventions: Dietary Supplement: Quorn Foods products
- Meat/fish products (Active Comparator)
  Interventions: Dietary Supplement: Meat/fish products

INTERVENTIONS:
Dietary Supplement: Quorn Foods products — 180 g mycoprotein (wet weight; corresponding to 45 g dry weight) per day (equates to approx. 215 g Quorn Foods products, depending on the product)
  Arms: Quorn Food products
Dietary Supplement: Meat/fish products — Standard meat/fish products matched to Quorn group for protein intake
  Arms: Meat/fish products

SUMMARY:
In overweight individuals (BMI > 27.5 kg/m2), does daily consumption of mycoprotein containing Quorn Food products lower blood cholesterol compared with daily meat/fish consumption?

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* BMI >27.5 kg/m2
* Non allergic to penicillin/mycoprotein
* Moderate levels of physical activity or below (self-identified; NDNS servey)
* Omnivores
* Not currently using cholesterol lowering medication

Exclusion Criteria:

* <18 or >70 years old
* BMI <27.5 kg/m2
* Allergies to penicillin/mycoprotein
* Heavy exercisers (self idenfiied)
* Vegetarian/vegans
* Currently using cholesterol lowering medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Postabsorptive blood cholesterol (free, total, LDL, HDL) concentrations | 4 weeks
  Test for intervention vs control differences in postabsorptive blood cholesterol levels (mMol) pre and post intervention

SECONDARY OUTCOMES:
Postprandial blood cholesterol concentration | 3 hours
  Test for intervention vs control differences in postprandial blood cholesterol levels (mMol) pre and post intervention
Fingerprick blood glucose concentration | 4 weeks
  Test for intervention vs control differences in blood glucose concentration (mMol) in postabsorptive and postprandial state
Satiety | 4 weeks
  Test for intervention vs control differences in satiety using a 10 centimetre 'Satiety Visual Analogue Scale' ratings, anchored by minimum to maximum response for a given aspect of satiety, where 0 cm is minimum and 10 cm is maximum
Hedonic visual analogue scale | 4 weeks
  Test for intervention vs control differences and changes in hedonic response using 10 cm 'Hedonic Visual Analogue Scale' ratings, anchored by minimum to maximum response for a given aspect of hedonic response, where 0 cm is minimum and 10 cm is maximum
Gastrointestinal side-effects | Once weekly, over 4 weeks
  Test for intervention vs control differences in tolerance of diet
Fingerprick blood c-peptide | 4 weeks
  Test for intervention vs control differences in C-peptide concentration (ng/ml) in postabsorptive and postprandial state
Fingerprick blood triglyceride concentration | 4 weeks
  Test for intervention vs control differences in blood triglyceride concentration (mMol) in postabsorptive and postprandial state

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Wall, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

REFERENCES:
- [Derived] Pavis GF, Iniesta RR, Roper H, Theobald HE, Derbyshire EJ, Finnigan TJA, Stephens FB, Wall BT. A four-week dietary intervention with mycoprotein-containing food products reduces serum cholesterol concentrations in community-dwelling, overweight adults: A randomised controlled trial. Clin Nutr. 2024 Mar;43(3):649-659. doi: 10.1016/j.clnu.2024.01.023. Epub 2024 Jan 24. PMID 38306892